CLINICAL TRIAL: NCT05823662
Title: Comparative Study Between DJ Stenting and Sildosin After Uretroscopic Lithotripsy for Lower Ureteric Stones
Brief Title: Double J Stenting and Sildosin After URSL for Lower Ureteric Stones
Acronym: DJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abou Elezz Abdel Fattah, Lecturer of Urology, Faculty of Medicine, Benha University, Benha, Egypt, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC 6-2-2023
Record Dates: First submitted 2023-03-16; First posted 2023-04-21 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Lower Ureteric Stones; Ureteroscopic Lithotripsy; DJ Stenting
MeSH Terms: interventions — silodosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DJ stent group (Experimental): A 5 Fr double J stent will be inserted and then removed after three weeks.
  Interventions: Procedure: DJ stent
- Silodosin group (Experimental): Patients will be given one capsule of silodosin 8 mg at the night for three weeks.
  Interventions: Drug: Silodosin

INTERVENTIONS:
Procedure: DJ stent — A 5 Fr DJ stent will be inserted and then removed after three weeks.
  Arms: DJ stent group
Drug: Silodosin — Patients will be given one capsule of silodosin 8 mg at the night for three weeks.
  Arms: Silodosin group

SUMMARY:
The aim of this prospective comparative clinical study to compare DJ stenting and Sildosin after ureteroscopic lithotripsy for lower ureteric stones.

DETAILED DESCRIPTION:
Ureteric calculi are known to affect approximately 10 - 15% of the overall population. The incidence of urolithiasis is rising over time. Most of these stones are known to pass spontaneously with or without expulsive medical therapy. The expulsion of calculus depends on the following factors: the calculus size and the location in the ureter (Alelign and Petros, 2018). The calculi expulsion rates change depending on these factors, with the expulsion rate ranging from 40% to 98% for calculi less than 5 mm. The calculi, which measure 6 mm or more have a spontaneous expulsion rate ranging between 35% to 50%.

Semirigid ureteroscopy (URS) lithotripsy has been shown to have high success rates for treating distal ureteric stones in many studies. However, URS is associated with some drawbacks, which may be risky and sometimes problematic.

The use of Double J (DJ) stent after ureteroscopy helps in the passage of residual fragments and prevents pain caused due to mucosal edema and obstruction. However, many patients complain of stent-related discomfort in the postoperative period. There is an additional need for stent removal, which is another surgical procedure adding to the cost of treatment. Despite its usefulness, the morbidity associated with these stents has been considered a potential health problem. However, many patients complain of stent-related discomfort in the postoperative period. There is an additional need for stent removal, which is another surgical procedure adding to the cost of treatment.

Silodosin is a highly selective alpha-1 adrenergic receptor antagonist which is used in the treatment of lower urinary tract symptoms (LUTS). Alpha-1 adrenergic receptors are densely found in the smooth muscle cells of the lower urinary tract, and silodosin relaxes them and improves the stent-related symptoms (SRS), and various studies have also shown similar effects. It has documented its use in the therapy of ureteric calculus.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 to 60 years,
* Diagnosed with lower ureteric stone and those patients willing to participate and follow up in the study.

Exclusion Criteria:

* Patients having a previous or present history of prostatic or bladder surgery, malignancy, neurological disorder, pelvic irradiation, and diabetes.
* Acute or chronic renal insufficiency, solitary kidney or congenital urinary abnormality, cardiac disease, postoperative residual stone fragments, multiple or bilateral ureteral stones, patients with bilateral stents or long-term stenting with frequent change of stents, history of interstitial cystitis, chronic cystitis or prostatitis.
* Medical treatment (α blockers, beta-blockers, calcium antagonists, 5 alfa reductase inhibitors, phosphodiesterase type 5 inhibitors, anticholinergics and cholinergic, nitrates).
* Pregnant and lactating women and patients not available for follow-up will be excluded from this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Stone-free rate | 3 weeks
  Stone free rate 24 hours and stone free rate 73 hours Stone free rate 73 hours Stone free rate 24 hours Stone free rate 73 hours Stone free rate will be recorded

SECONDARY OUTCOMES:
Operative time | Intraoperatively
  Operative time in minutes will be recorded
Comlications | 24 hours Postoperative
  Complications as fever, flank pain, Lower Urinary lower urinary tract Symptoms or hematuria

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospitals, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study will be available under a reasonable request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: One year after the end of the study